CLINICAL TRIAL: NCT00197314
Title: A Randomized Controlled Trial of Circular Muscle Exercises (Paula Method) vs. Pelvic Floor Training (Kegel Exercises) for Urinary Stress Incontinence in Women
Brief Title: Effectiveness of Circular Muscle Exercise (Paula Method) Versus Kegel Exercise for Urinary Stress Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0204-20-22-HMO-CTIL
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2005-09

CONDITIONS: Urinary Stress Incontinence (SI)
Keywords: Urinary stress incontinence; Randomized trial; circular muscle training; pelvic floor training; bioequivalence
MeSH Terms: conditions — Urinary Incontinence, Stress

INTERVENTIONS:
Behavioral: circular muscle exercises versus pelvic floor exercises

SUMMARY:
This is a randomized controlled trial comparing two methods of exercise for the treatment of stress incontinence ( loss of urine after physical exertion) in women. We are comparing the Paula method of circular muscle exercise, in which circular muscles controlling sphincters of the body (such as the eyes, mouth and rectum) are exercised, with pelvic floor training (Kegel exercises) in women in the community. The study hypothesis is that the effectiveness of circular muscle exercises is equivalent to pelvic floor training among women with this disorder.

DETAILED DESCRIPTION:
Background: Urinary stress incontinence(SI) is defined as involuntary urinary loss which appears during increased intra-abdominal pressure which can be measured objectively. It is an important social and hygienic problem. Its prevalence varies fron 12-55% depending on age, and geography. The economic costs of this condition were estimated to reach 24 billion dollars in the US in 1995. The objectives of this study are to evaluate two non-invasive methods of treatment of stress incontinence.

Methods: 200 women who chosen from the community and suffering from SI will enter the study and will be randomized to one of two arms. The first arm is the Paula method of circular muscle exercises: these women will receive private lessons from a registered Paula instructor. The system is based on activating circular muscles in the body. The second arm will receive instruction in pelvic floor muscle training by a physiotherapist.

The clinical trial will compare the efficacy of the methods for the treatment of SI. The candidates for inclusion in the trial will undergo a gynecological exam and a "Pad Test". The efficacy will be measured in terms of changes in the Pad test (quantity of urinary leakage) and subjective reports of the participants on leakage, quality of life and sexual function.

ELIGIBILITY:
Inclusion Criteria:ambulatory women, aged 20-65, living in Jerusalem area, able to understand instruction in Hebrew or English, suffering from urinary stress incontinence with a positive Pad test of at least 1 gm -

Exclusion Criteria:pregnant,within 12 weeks of delivery,6 weeks since abortion,breastfeeding, illnesses which limit physical activity (cardiac, respiratory, psychiatric and neurological), Pad test < 1gm,pelvic surgery within last 6 months, genital prolapse Grade 3 or higher, previous surgery for urinary incontinence, previous pelvic radiation therapy

-

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-06; Study Completion 2006-03

PRIMARY OUTCOMES:
Mean change in grams of urinary leakage as measured by Pad test

SECONDARY OUTCOMES:
Quality of life as measured by IQOL scale, sexuality as measured by questionnaire, subjective assessment of SI and general health

CONTACTS AND LOCATIONS:
Overall Officials: Ora B Paltiel, MD, Principal Investigator — Hadassah University Hospital
Locations (1):
- Dr. Ora Paltiel, Jerusalem, Israel

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322